CLINICAL TRIAL: NCT02697370
Title: Efficacy and Cost Effectiveness of Standard Versus Pharmacokinetic Dosing During Factor VIII Prophylaxis in Adult Patients With Severe Haemophilia A
Brief Title: Efficacy and Cost Effectiveness of Pharmacokinetic Dosing in Haemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Collaborators: University of Wales Cardiff United Kingdom (UK) (Unknown); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/SC/0363
Record Dates: First submitted 2016-02-18; First posted 2016-03-03 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Severe Haemophilia A
Keywords: Haemophilia A prophylaxis pharmacokinetic dosing
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pharmacokinetic based factor VIII dosage (Other): Patient's routine prophylactic factor VIII concentrate infusion will be given in the morning and the exact time (hours and minutes) and dose recorded. There is no wash out so the date, time and dose of the previous 2 prophylactic doses must be accurately known. Samples will be collected that afternoon, the following morning and the following afternoon. Samples can be taken at any convenient time but the exact time must be recorded. Factor VIII levels will be measured and this pharmacokinetic data will be used to calculate the dose of factor VIII (to be infused on alternate days) required to maintain a predicted factor VIII ≥1.5 IU/dL at all times(this will be rounded up to the nearest full 250 IU vial)
  Interventions: Drug: Pharmacokinetic based dosage change

INTERVENTIONS:
Drug: Pharmacokinetic based dosage change — Pharmacokinetic based dosing of factor VIII prophylaxis treatment compared to standard prophylactic regimens based on weight.Prophylaxis is prescribed according to routine clinical practice with prophylaxis prescribed on alternate days to maintain predicted target trough of ≥1.5 IU/dL based on sparse blood sampling and Bayesian pharmacokinetic estimation
  Other Names: Factor VIII replacement therapy - non brand specific

SUMMARY:
Patients with severe Haemophilia A need prophylactic factor VIII to reduce their risk of joint and soft tissue bleeds and to prevent or reduce joint damage. It is common practice to give enough factor VIII to maintain the trough level above 1% of normal and this has been supported in retrospective studies.

The amount of factor VIII required to maintain this trough level varies markedly between patients because their factor VIII half lives are different. This study will assess the role of regular pharmacokinetic (PK)monitoring and dose adjusted factor VIII to establish whether this is a more cost effective way of giving treatment and whether it is feasible in routine clinical practice. Patients will be treated for 6 months with their standard factor VIII regimen and followed up to establish their bleed frequency. They will then receive pharmacokinetic adjusted factor VIII to maintain a trough above 1.5% for a year and their bleed rate compared to standard treatment. If they have increased break through bleeds their factor VIII will be increased to maintain a trough of 3%.

DETAILED DESCRIPTION:
Study procedures

Recruitment and Consent Patients with severe Haemophilia A who are taking any regular prophylactic regimen with infusions of factor VIII at least 3 times a week and do not have a target joint will be eligible. Initial approach will be made by the Principal Investigator at the patients next scheduled review appointment.

Phase 1: Study enrolment Participants will be allocated a unique patient number upon enrolment into the study.

The following will be recorded at study enrolment:

* Date of birth
* Height and weight
* Baseline factor VIII based on historical data from the patient record
* History of a factor VIII inhibitor
* Information on the number and site of haemarthroses and soft tissue bleeds and total amount of factor VIII used in the preceding 12 months will be recorded, if known
* Quality of life assessment by Utility-EQ5D
* Joint assessment by Haemophilia Joint Health Score (HJHS)

An abbreviated (3 sample) pharmacokinetic study will be undertaken as follows:

There will be no wash out. The patient's routine prophylactic infusion will be given in the morning and the exact time (hours and minutes) and dose recorded. Since there is no wash out the date, exact time and dose of the previous 2 prophylactic doses (i.e. 3 infusions in total) must be accurately known.

Blood samples will then be taken to measure

1. Factor VIII levels
2. Von Willebrand factor (VWF) antigen level
3. Von Willebrand factor propeptide
4. Von Willebrand factor: factor VIII binding
5. Coagulation screen
6. Inhibitor assay by Nijmegen modification of Bethesda assay & ELISA (only first afternoon timepoint)
7. CRP (only first afternoon time point)

Samples for above tests will be collected that afternoon, the following morning and the following afternoon. The samples can be taken at any convenient time but the exact time (hours and minutes) must be recorded. Factor VIII levels will be measured. The patient's weight (kg), amount and exact time of the last 3 factor VIII infusions, measured factor VIII levels and exact times of when the samples were taken will be communicated to the centre in Uppsala and the pharmacokinetic parameters established using a Bayesian procedure based on a population model.

The following will be established or recorded from the notes if already known

1. Blood group
2. Factor VIII mutation
3. DNA testing other genes that may affect factor VIII clearance e.g. lipoprotein receptor
4. Factor VIII and Von Willebrand factor genetic sequence

Phase 2: Standard treatment for 6 months

The patients will remain on their routine prophylactic regimen as determined by their clinician for a period of 6 months. The patient's current factor VIII product will be used and the factor VIII product should not change throughout the study. Patients will be instructed to give all prophylactic infusions in the morning (defined as before midday).

The following procedures will be undertaken:

Patients will keep a diary of:

a All factor VIII infusions. Information will be collected on the dose of factor VIII, time(hours and minutes) of infusion and reason for infusion (prophylaxis or treatment of a bleed).

b Bleeding events. Information will be collected on the type of bleed (haemarthrosis or soft tissue), site (identified by specific joint or position), cause (atraumatic or traumatic with precipitating event), symptoms or signs of swelling, pain or loss of function and time.

Every 2 weeks for the first 2 months and subsequently monthly a nurse or doctor will make contact by telephone, email or text to confirm that the diary is being completed.

At 3 months a doctor will review the patient and the diary and make appropriate changes to treatment. Patients will have open access to contact or attend the Haemophilia Centre as is currently the case. The clinician will make appropriate changes to treatment.

Phase 3: Pharmacokinetic tailored treatment

At the end of phase 2, i.e. 6 months after the start of the study the patient will attend the haemophilia centre for:

* Review of bleed chart diary and treatment
* QOL assessment (Utility-EQ5D)
* Joint assessment (HJHS)
* An abbreviated (3 sample) pharmacokinetic study will be undertaken as follows:

As before there will be no wash out. The patient's routine prophylactic infusion will be given in the morning and the exact time and dose recorded. Also the date, exact time and dose of the previous 2 prophylactic doses (i.e. 3 infusions in total) must be accurately known and recorded.

Blood samples will then be collected to measure parameters as in Phase 1

The centre in Uppsala will use the pharmacokinetic data to calculate the dose of factor VIII (to be infused on alternate days) required to maintain a predicted factor VIII ≥1.5 IU/dL at all times, and inform the patient's centre of the dose to prescribe (this will be rounded up to the nearest full 250 IU vial).

This regimen will be prescribed for 12 months i.e. months 7-18 of the study. The patient's current factor VIII product will be used. Patients will be instructed to give all prophylactic infusions in the morning (defined as before midday).

The patients will follow the same procedures and keep a diary as in Phase 1.

At 3, 6 and 9 months (+/- 2 weeks) of starting the pharmacokinetic tailored treatment phase (i.e. at the end of 9, 12 and 15 months (+/- 2 weeks) from starting the study), a doctor will review the patient and the diary and make appropriate changes to treatment according to the Phase 3 dose escalation protocol. At each of these visits participants will have their weight and factor VIII levels measured As before there will be no wash out. The patient's routine prophylactic infusion will be given in the morning and the exact time and dose recorded. The date, exact time and dose of the previous 2 prophylactic doses must also be accurately known and recorded.

Blood samples will be collected that afternoon, the following morning and the following afternoon and parameters measured as in Phase 1.

The Uppsala centre will calculate the pharmacokinetic parameters. Based on these results the dose required by the patient will be reviewed and recommend the most appropriate dose to maintain a trough level ≥ 1.5 IU/dL.

Dose escalation Phase 2

If a participant experiences more than one clinically significant bleed in a 4 month period during phase 2 (clinician routine prescribing) treatment will be adjusted by the clinician according to that clinician's routine practice. This could mean that the prophylactic dose does not change.

Phase 3

If a participant experiences more than one clinically significant bleed in a 4 month period during phase 3 (pharmacokinetic tailored dosing) a dose escalation will occur. The participant will have their prophylaxis dose increased to sustain a trough factor VIII level above 3 IU/dL i.e. the prophylactic dose will be doubled. If the participant has more than one clinically significant bleed in a subsequent 4 month period they will be withdrawn from the study and return to routine care.

This means that no more than 4 clinically significant bleeds, per participant, will be permitted in phase 3 (1 year) of the study. This figure is based on the finding that 5% of patients on full dose standard prophylaxis have more than 3 bleeds per year and that the median number of bleeds in prospective prophylaxis studies in adult patients is between 0 and 3 per year.

Study end

After 18 months the patients will undergo:

* Weight measurement
* Diary review of bleeds, treatments and adverse events
* Quality of life assessment by Utility-EQ5D
* Joint assessment by HJHS
* Blood will be taken for parameters as in Phase 1

The patient will then exit the study.

Adverse Events

A clinical review will be held after each clinically significant bleed on phase 3 of the study. If a participant experiences more than 4 bleeds during phase 3 of the study, this will be classed as an adverse event and the participant will be withdrawn from the study. If more than 5 participants have more than 1 spontaneous clinically significant bleed in a 4 month period after the dose escalation to 3%, the study will be reviewed by the IDMC and if confirmed all participants will be reverted back to standard care and the study terminated.

Pharmacokinetic analysis and dose recommendation

Calculation of pharmacokinetic parameters and the dose of factor VIII for prophylactic during phase 3 will be performed at the Department of Pharmaceutical Biosciences, Uppsala University, under the supervision of Professor Bjorkman using NonmemR software. The factor VIII levels, time and dose of factor VIII infusions and patients' weight will be sent to Uppsala. No other information will be sent. The dose recommendation will be sent to the treating centre by secure email within 7 days. The local centre will use the same information available to Uppsala and the TCIworksR software to calculate the patients' pharmacokinetics and dose recommendations. The dose recommendation of Uppsala will be used if the local recommendation is different.

Method for measurement of patient pharmacokinetics

The study patients' pharmacokinetic parameters will be estimated by a Bayesian procedure based on a population model, according to methods already in use e.g. for aminoglycoside antibiotics, digoxin or immunomodulating drugs. Pharmacokinetic parameter estimates will be obtained from the 6 month results and then be updated when new data is obtained after 9, 12, 15 and 18 months. A complete population pharmacokinetic analysis will be performed after collection of all data with the aim to investigate:

1. Intra-individual (inter-occasion) variance in pharmacokinetics in relationship to inter-individual variance.
2. The relationship of pharmacokinetic variables with patient characteristics (as determined at each study occasion), in particular VWF:Ag level, VWF:factor VIII binding, VWF propeptide, blood group, inflammation (CRP), inhibitor titre and factor VIII mutation.

Analysis

First; the primary and secondary endpoints will be compared between phase I and II i.e. number of clinically significant bleeds, total bleeds, clotting factor consumption/kg, quality of life, and joint status. These comparisons will be performed using paired T-tests and non parametric tests.

Second; the performance of pharmacokinetic calculation methods will be assessed: predicted FVIII levels will be compared to measured FVIII levels, and inter- as well as inter patient variability of PK parameters will be assessed.

Third; the determinants of bleed rate will be addressed using multivariate regression with a negative binomial model and joint bleeds as well as total bleeds as the outcome. Using this approach, the independent effects of calculated weekly time below 1%, baseline arthropathy, and physical activity will be assessed.

Fourth; the association of patient characteristics (age, weight, BMI, blood group, VWF level, factor VIII mutation, VWF:FVIII binding, VWF polymorphisms, current or past history of factor VIII inhibitor or inflammation) and PK parameters (AUC and half life) will be assessed using multivariate regression techniques.

Finally, patient characteristics associated with treatment failure (e.g. lower than predicted factor VIII levels, higher activity, non-reproducible pharmacokinetic results or lack of adherence) will be assessed, using descriptive statistics and multivariate logistic regression if possible.

The study will be deemed to have a positive outcome if:

1. Patients are treated with factor VIII doses calculated from individual pharmacokinetics for 12 months in at least 80% of cases.
2. The median increase in clinically significant bleeds in the pharmacokinetic dosed arm compared to routine practice is less than 2 in 80% of the patients
3. There is a statistically significant reduction in the average factor VIII usage in the pharmacokinetic dosed period compared to the clinician dosed period.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A (baseline factor VIII < 1IU/dL)
* Age 18 years and above
* Patients taking any regular prophylactic regimen (defined as regular factor VIII infusions, at least 3 times a week, with the aim minimising haemarthroses and other clinically significant bleeds).
* Low titre inhibitors, past history of an inhibitor, abnormal liver function, drugs that interfere with haemostasis and low CD4 counts are allowed.

Exclusion Criteria:

* Presence of a target joint on prophylaxis (defined as 3 bleeds into one joint, during a 6 month period,during the last year).
* The occurrence of more than 3 haemarthroses in the last year which required more than 2 infusions to resolve

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The number of clinically significant bleeds in patients taking routine prophylaxis compared to prophylaxis dosed according to individual pharmacokinetics | 18 months
  Factor VIII dosage tailored treatment based on pharmacokinetics

SECONDARY OUTCOMES:
Compare the factor VIII usage between the two regimens | 18 months
Compare the total number of all haemarthroses between the two regimens | 18 months
Compare the total number of all soft tissue bleeds between the two regimens | 18 months
Compare the quality of life (EQ5D) between the two regimens | 18 months
Compare the patients' joint status between the two regimens using the HJHS score. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Savita Rangarajan, FRCP FRCPath, Principal Investigator — Basingstoke & North Hampshire Hospital
Locations (1):
- Basingstoke & North Hampshire Hospital, Basingstoke, United Kingdom